CLINICAL TRIAL: NCT03769831
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR2285 Tablets in Healthy Subjects
Brief Title: The PK/PD Study of SHR2285 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SHR2285-101
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2018-12

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR2285 (Experimental): Up to 7 cohorts of healthy subjects will receive a single dose of oral SHR2285 tablet.
  Interventions: Drug: SHR2285
- Placebo (Experimental): Up to 7 cohorts of healthy subjects will receive a single dose of oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR2285 — Ascending dose oral adminstration
  Arms: SHR2285
Drug: Placebo — Ascending dose oral adminstration
  Arms: Placebo

SUMMARY:
Thrombosis is a maladaptive process of vascular occlusion and remains a primary cause of cardiovascular morbidity and mortality, The dose-limiting issue with available anticoagulant therapies is bleeding. The primary objective of this study is to assess the safety and tolerability of SHR2285 tablets in healthy subjects. In addition, this study will provide information on Pharmacokinetics and Pharmacodynamics of SHR2285 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18-45
2. subjects with no cardiovascular disease, sitting blood pressure: 90mmHg ≤SBP<140mmHg and 50mmHg ≤DBP<90mmHg;
3. body mass index (BMI) between 18 to 28, and a total body weight: male ≥50.0 kg and <90.0 kg; female ≥45.0 kg and <90.0 kg
4. Participant in general good health. No clinically significant findings in laboratory parameters or clinically significant abnormality on X-ray

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin > 1X ULN during screening/baseline;
2. Abnormal coagulation function;
3. A clinical history of coagulation dysfunction；subjects with adverse reaction of antiplatelet drugs or anticoagulant drugs.
4. Subjects with severe trauma or surgery within 3 months prior to the screening；
5. Known blood donation within 30 days pre-dose; donating≥400 ml of blood 3 months pre-dose;
6. Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive;
7. 3 months prior to screening involved in any drug or medical device clinical subjects, or within 5 half-life of drugs before screening;
8. Pregnant or Serum β-hCG > 5mIU/mL at baseline or women who are breastfeeding; etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events | Pre-dose to 7 days after dose administration

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SHR2285 | Pre-dose to 2 days after dose administration
Maximum observed serum concentration (Cmax) of SHR2285 | Pre-dose to 2 days after dose administration
Time to maximum observed serum concentration (Tmax) of SHR2285 | Pre-dose to 2 days after dose administration
Time to elimination half-life (T1/2) of SHR2285 | Pre-dose to 2 days after dose administration
Apparent total clearance of the drug from plasma after oral administration(CL/F) of SHR2285 | Pre-dose to 2 days after dose administration
Apparent volume of distribution after non-intravenous administration (V/F) of SHR2285 | Pre-dose to 2 days after dose administration
Mean Residence Time(MRT) of SHR2285 | Pre-dose to 2 days after dose administration
Change of APTT, PT, INR from baseline. | during Pre and Post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen R, Guan X, Hu P, Dong Y, Zhu Y, Zhang T, Zou J, Zhang S. First-In-Human Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of SHR2285, a Small-Molecule Factor XIa Inhibitor in Healthy Subjects. Front Pharmacol. 2022 Feb 10;13:821363. doi: 10.3389/fphar.2022.821363. eCollection 2022. PMID 35222036